CLINICAL TRIAL: NCT03030339
Title: Vitamin A Status and Risk of Excessive Vitamin A Intake Among Urban Filipino Children Exposed to Multiple Vitamin A Intervention Programs
Brief Title: Vitamin A Status and Risk of Excessive Vitamin A Intake Among Urban Filipino Children
Acronym: GloVitAS-P
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Newcastle University (Other); Penn State University (Other); Helen Keller International (Other); Food and Nutrition Research Institute, Philippines (Other Government); Global Alliance for Improved Nutrition (Other); Bill and Melinda Gates Foundation (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: 903681; OPP1115464 (Other Grant/Funding Number: Other)
Record Dates: First submitted 2017-01-17; First posted 2017-01-25 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Vitamin A Status
Keywords: Vitamin A status; infant; dietary assessment; retinol isotope dilution; breast milk intake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, red and white cells, dried blood spots, breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: High VA intake, recent VAS: Children who are exposed to multiple vitamin A (VA) programs, have received a high-dose VA supplement (VAS; 200,000 IU) in the past month, and are identified as being likely to have chronic excessive dietary VA intake
  Interventions: Other: High VA intake, recent VAS
- Group 2: High VA intake: Children who are exposed to multiple vitamin A (VA) programs, have received a high-dose VA supplement (200,000 IU) in the past 3-6 months, and are identified as being likely to have chronic excessive dietary VA intake.
  Interventions: Other: High VA intake
- Group 3: Low/adequate VA intake: Children who are not exposed to multiple vitamin A (VA) programs, have received a high-dose VA supplement in the past 3-6 months, and are identified as being likely to have chronic low to adequate dietary VA intake.
  Interventions: Other: Low/adequate VA intake

INTERVENTIONS:
Other: High VA intake, recent VAS — Children who are exposed to multiple VA programs, have received a high-dose VA supplement (VAS; 200,000 IU) in the past month, and are identified as being likely to have chronic excessive dietary VA intake.
  Groups: Group 1: High VA intake, recent VAS
Other: High VA intake — Children who are exposed to multiple VA programs, have received a high-dose VA supplement (200,000 IU) in the past 3-6 months, and are identified as being likely to have chronic excessive dietary VA intake.
  Groups: Group 2: High VA intake
Other: Low/adequate VA intake — Children who are not exposed to multiple VA programs, have received a high-dose VA supplement in the past 3-6 months, and are identified as being likely to have chronic low to adequate dietary VA intake.
  Groups: Group 3: Low/adequate VA intake

SUMMARY:
The goal of this study is to assess whether children 12-18 months of age who are exposed to multiple large-scale vitamin A programs, and who are likely to have vitamin A intakes above the tolerable upper intake level (UL), have higher total body vitamin A stores and biomarkers of excessive vitamin A status, compared to children 12-18 months of age who have adequate vitamin A intake.

DETAILED DESCRIPTION:
This is an observational study with 3 groups, which are identified using a screening tool to obtain information on exposure to vitamin A programs and consumption of vitamin A-rich foods and supplements. Children and their mothers are studied over the course of one month to determine 1) child total body vitamin A stores, using the 13C retinol isotope dilution method, 2) the child's vitamin A intake, using multiple dietary assessment methods, 3) total breast milk intake (among breastfeeding children), using the dose-to-mother deuterium dilution method, and 4) potential biomarkers of excessive vitamin A status, including markers of bone and liver health. Blood collection is structured in a "Super-Child" design, to construct plasma retinol kinetic curves. Other indicators related to vitamin A nutrition among children will be measured, in addition to the vitamin A intake and breast milk vitamin A concentration (for breastfeeding mothers) of the mother.

ELIGIBILITY:
Inclusion Criteria:

* Children 12-18 months of age, and their mothers (18-49 years of age)
* Living in selected communities in the National Capital Region of the Philippines
* The mother and child must plan to stay in the study area for the duration of the study.
* Child's estimated vitamin A intake and exposure to vitamin A programs must meet eligibility criteria for one of three groups, based on a screening questionnaire administered by an interviewer to the child's mother.

Eligibility criteria for children in Group 1: 1) consumed MNP or a multi-vitamin preparation that contains vitamin A in the previous 7 days, 2) consumed at least one fortified staple food (oil or wheat flour) in the previous 7 days, 3) consumed breast milk or fortified milk in the past 24 hours, 4) received a high-dose VA capsule during the previous month, and 5) received a screening tool 'score' suggesting VA intake above 600 µg retinol/d.

Eligibility criteria for children in Group 2: will include children who: 1) consumed MNP or a multi-vitamin A preparation that contains vitamin A in the previous 7 days, 2) consumed at least one fortified staple food (oil or wheat flour) in the previous 7 days, 3) consumed breast milk or fortified milk in the past 24 hours, 4) received a high-dose VA capsule in the previous 3-6 months, and 5) received a screening tool 'score' suggesting VA intake above 600 µg retinol/d.

Eligibility criteria for children in Group 3: will include children who: 1) received a high dose VA capsule during the previous 3-6 months, and 2) received a screening tool 'score' suggesting VA intake 200-500 µg/d.

Exclusion Criteria:

* The child did not receive a high-dose VA capsule during the most recent national campaign
* The mother or child has chronic disease
* The child has moderate or severe anemia (Hb <10 g/dL)
* The mother or child has signs or symptoms of vitamin A deficiency (Bitot's spots, conjunctival xerosis, nightblindness)
* The child has weight for length < -2 z-scores of the median of the WHO growth standards
* The mother is breastfeeding more than one child

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 12-18 months of age and their mothers in selected neighborhoods in the National Capital Region of the Philippines
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Total body vitamin A stores among children 12-18 mo of age | 28-day study period
  Estimated using the 13C-retinol dilution method
Total dietary vitamin A intake among children 12-18 mo of age | 28-day study period
  Estimated using 24-hour dietary recalls, observed weighed food records, food and supplement frequency questionnaire, breast milk vitamin A concentration, and total breast milk intake (measured by the dose-to-mother deuterium dilution technique)
Total breast milk intake (among breastfeeding children 12-18 mo of age) | 15-day study period
  Estimating using the dose-to-mother deuterium dilution technique.

SECONDARY OUTCOMES:
Plasma or serum retinol among children 12-18 mo of age | 28-day study period
Plasma or serum retinol-binding protein among children 12-18 mo of age | 28-day study period
Ratio of retinol to retinol-binding protein among children 12-18 mo of age | 28-day study period
Retinol metabolites among children 12-18 mo of age | 28-day study period
Transthyretin among children 12-18 mo of age | 28-day study period
Bone health markers among children 12-18 mo of age | 28-day study period
Liver function markers among children 12-18 mo of age | 28-day study period
Consumption of fortifiable foods among women | 28 day study period
  Estimated by combining data from 24-hour recalls, observed weighed food records, food frequency questionnaires, and the Fortification Assessment Coverage Tool
Consumption of fortifiable foods among children | 28 day study period
  Estimated by combining data from 24-hour recalls, observed weighed food records, food frequency questionnaires, and the Fortification Assessment Coverage Tool
Total vitamin A intake among women | 28-day study period
  Estimated using 24-hour dietary recalls and food frequency questionnaires
Breast milk vitamin A concentration among lactating women | 28-day study period

OTHER OUTCOMES:
Total food and nutrient intakes among women | 28-day study period and 30 days prior to study period
Total food and nutrient intakes among children | 28-day study period and 30 days prior to study period
Infant weight-for-length z score | At recruitment
Infant length-for-age z score | At recruitment
Systemic inflammation among children | 28-day study period
Iron status among children | 28-day study period
Zinc status among children | 28-day study period
Hepatitis infection among children | 28-day study period
Genetic markers related to vitamin A metabolism among children | 28-day study period
Infant hemoglobin concentration | At enrollment
Infant morbidity symptoms | 28-day study period and previous 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lietz, Study Director — Newcastle University
Locations (1):
- Block 37 Health Center, Mandaluyong, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.

REFERENCES:
- [Derived] Engle-Stone R, Miller JC, Reario MFD, Arnold CD, Stormer A, Lafuente E, Oxley A, Capanzana MV, Cabanilla CVD, Ford JL, Clark A, Velavan TP, Brown KH, Lietz G, Haskell MJ. Filipino Children with High Usual Vitamin A Intakes and Exposure to Multiple Sources of Vitamin A Have Elevated Total Body Stores of Vitamin A But Do Not Show Clear Evidence of Vitamin A Toxicity. Curr Dev Nutr. 2022 Jul 25;6(8):nzac115. doi: 10.1093/cdn/nzac115. eCollection 2022 Aug. PMID 36060221
- [Derived] Oxley A, Engle-Stone R, Miller JC, Reario MFD, Stormer A, Capanzana MV, Cabanilla CVD, Haskell MJ, Lietz G. Determination of Vitamin A Total Body Stores in Children from Dried Serum Spots: Application in a Low- and Middle-Income Country Community Setting. J Nutr. 2021 May 11;151(5):1341-1346. doi: 10.1093/jn/nxaa446. PMID 33755155
- [Derived] Ford JL, Green JB, Haskell MJ, Ahmad SM, Mazariegos Cordero DI, Oxley A, Engle-Stone R, Lietz G, Green MH. Use of Model-Based Compartmental Analysis and a Super-Child Design to Study Whole-Body Retinol Kinetics and Vitamin A Total Body Stores in Children from 3 Lower-Income Countries. J Nutr. 2020 Feb 1;150(2):411-418. doi: 10.1093/jn/nxz225. PMID 31535129